CLINICAL TRIAL: NCT06602336
Title: A Single Centre Study Comparing Continuous Interstitial Fluid Lactate Detection (as Measured by Change in Current) to Standard Measurements of Change in Venous and Arterial Lactate in Patients Undergoing Elective Coronary Artery Bypass Graft Surgery and/or Valve Replacement.
Brief Title: A Single Centre Study Comparing Continuous Interstitial Fluid Lactate Detection to Standard Measurements of Lactate in Patients Undergoing Elective Coronary Artery Bypass Graft Surgery and/or Valve Replacement.
Acronym: CONTINUUM LINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 346076
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Bypass; Coronary Artery Bypass Graft; Coronary Artery Bypass Graft Surgery (CABG); Valve Replacement; Valve Surgery; Cardiovascular; CABG
Keywords: device; cardiovascular; coronary artery bypass surgery; replacement valve surgery; Continuous lactate monitor; CABG; wearable device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Lactate Device (Experimental): Continuous interstitial fluid lactate monitoring using the Abbott Investigational Lactate Device
  Interventions: Device: Continuous Lactate Monitoring Device

INTERVENTIONS:
Device: Continuous Lactate Monitoring Device — Continuous interstitial fluid lactate monitoring using the Abbott Investigational Lactate Device.

SUMMARY:
The main goal of this study is to see if a wearable device can reliably track changes in lactate levels in the body. We'll compare the device's readings to standard blood tests to ensure accuracy. If successful, this device could reduce the need for frequent blood tests during surgery recovery, making patients more comfortable. It might also be useful in emergency rooms for quick diagnoses, especially for patients with chest pain.

This study will take place at Barts Hospital with patients having planned coronary artery bypass graft (CABG) and/or replacement valve surgery. Participants will wear the sensors on their upper arm, during which the sensors will continuously measure lactate levels. Participants will also have hourly blood samples taken.

In the future, the data from this new device will be used to train computer algorithms to provide quick responses that help manage a patient's condition, improving future medical care and technology.

DETAILED DESCRIPTION:
Summary of the study design and methodology

The research nurse or doctor will meet with the patient to explain the study and check the following:

Pre-screening: The research nurse, who may also be part of the patient's direct care team, will look at the records for patients who are attending St Bartholomew's hospital for cardiac surgery for grafts and/or valve replacement.

Informed Consent: If the patient is eligible, and would like to take part in the study, the research nurse or doctor will ask the patient to sign a consent form indicating their willingness to participate in the study.

Screening: The research nurse or doctor will collect demographic information from the patient and ensure the patient meets the study's inclusion and exclusion criteria.

Sensor Application: Up to 5 days pre-surgery, the research nurse will place two lactate sensors on the patient's arm. The sensor has a 24 hour warm-up period prior to continuously measuring the patient's lactate levels.

Pre-Surgery Admission: The research nurse will gather details about the patient's medical history and current medications. The patient will have their blood pressure, heart rate, respiratory rate, weight, and height measured, and an ECG performed. Baseline blood samples will be collected as per the standard of care pre-CABG and/or valve surgery.

CABG and/or replacement valve surgery: The patient will then undergo their planned CABG and/or replacement valve surgery as usual.

Blood Sampling: The patient will have hourly blood samples taken through the tubes inserted for their surgery for up to 14 hours to compare with the sensor readings. These samples will include 12 arterial lactate, 12 central venous lactate, and 12 venous troponin samples. Hourly measurements of the patient's blood pressure, heart rate, and respiratory rate will be taken, and any medication changes will be noted.

Sensor Removal: Up to 48 hours post-surgery, the sensors will be removed, and the patient's skin will be checked for any changes, like a rash. The patient will also have their blood pressure, heart rate, and respiratory rate measured, and an ECG performed. Any changes to the patient's medication will be noted.

Follow-Up: The study team will monitor the patient for up to 24 hours after the sensor is removed or until the patient is discharged from the hospital (whichever is earlier). The study team will note any medication changes, measure the patient's blood pressure, heart rate, and respiratory rate, and perform an ECG.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* ≥18 to ≤ 90 years old
* Successful surgery as defined by the below criteria (which will be recorded in the eCRF):

  * Operative Success: The successful completion of coronary artery bypass grafting (CABG) and/or valve insertion with grafts and/or valves
  * Absence of the following complications:
  * Significant bleeding requiring reoperation
  * Evidence of major life-changing stroke

Exclusion Criteria:

* Previous coronary artery bypass grafting
* Recent acute coronary syndrome (within 4 weeks of planned consent date)
* Heart failure with EF less than 35% (from TTE or CT from past 6 months - if both available lower value will be used).
* Chronic severe renal failure (estimated eGFR less than 30 mL/min/1.73m2 by the MDRD formula recorded at time of consent)
* Severe anaemia (Hb less than 10 recorded at time of consent)
* Known or suspected allergies to medical grade silicone adhesives
* Pre-existing skin condition on the upper arm where the device would be applied, including recent burns/ scalds, open wounds or clinically significant skin lesions.
* Patients with implanted medical devices such as pacemakers or other CLMs
* Severe liver cirrhosis (≥ stage III)
* Lymphoedema or pitting oedema at the time of consent
* Pregnancy
* History of ongoing malignant disease
* Hypoalbuminaemia (less than 35 g/L recorded at time of consent)
* Those lacking capacity to consent or are deemed vulnerable adults
* Unable to speak English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Continuous lactate sensor measurement compared venous and arterial blood gas lactate measurements. | 14 hours
  Correlation coefficients describing the strength of association between the electrical signal from the continuous interstitial fluid lactate measurements and laboratory lactate measurements. Evaluate the change in interstitial fluid lactate measurements via a surrogate output of change in current (nA; using an investigational device by Abbott Diabetes Care Ltd.) to local Radiometer ABL 90 venous and arterial blood gas lactate measurements measured hourly up to 12 samples within a 14-hour period post-elective CABG/valve replacement surgery.
Continuous lactate sensor measurement compared Troponin-T | 14 hours
  Correlation coefficients describing the strength of association between the electrical signal from the continuous interstitial fluid lactate measurements and venous laboratory measurements of high-sensitivity troponin-T. Evaluate the relationship between the current (nA) output of a continuous interstitial fluid lactate monitor (using an investigational device by Abbott Diabetes Care Ltd.) and venous laboratory measurements of high-sensitivity troponin-T measured hourly up to 12 samples within a 14-hour period post-elective CABG/valve replacement surgery.

SECONDARY OUTCOMES:
Relationship between arterial and venous lactate measurements | 14 hours
  Correlation coefficients describing the strength of association between arterial and central venous lactate measurements measured hourly up to 12 samples within a 14- hour period post-elective CABG and/or valve replacement surgery.
Relationship between arterial and venous lactate and venous troponin measurements | 14 hours
  Correlation coefficients describing the strength of association between arterial and central venous lactate and venous troponin measured hourly up to 12 samples within a 14-hour period post-elective CABG and/or valve replacement surgery.
Functionality of the device for up to 48 hours post-surgery. | 48 hours
  Proportion of devices that are able to give a continuous electrical signal for the duration of use post-surgery.
Evaluate safety of lactate sensor | Up to 8 days
  Number of patients experiencing adverse reactions or serious adverse reactions to the lactate investigational device.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anthony Mathur, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided